CLINICAL TRIAL: NCT06531057
Title: Determination Of Factors Affecting Mobility In Patients Undergoing Abdominal Surgery
Brief Title: Determination Of Factors Affecting Mobility
Status: Completed | Type: Observational
Sponsor: Sanko University (Other)
Responsible Party: Principal Investigator, Ebru Karaaslan, research assistant, Sanko University
Other Study IDs: SankoU-Nursing-EK-003
Record Dates: First submitted 2024-07-28; First posted 2024-07-31 (Actual); Last update posted 2024-08-05 (Actual); Status verified 2024-08

CONDITIONS: Surgery
Keywords: postoperative care; Mobilization; Surgical Nursing

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- cross sectional: The population of the study consisted of 236 patients who underwent cholecystectomy, appendectomy, hernia surgery and bariatric surgery in the general surgery clinic of the specified hospital on the dates of data collection. Among these patients, 152 patients who met the sampling criteria and volunteered to participate in the study were included in the sample.

SUMMARY:
This descriptive study was conducted to determine the factors affecting mobility in patients undergoing abdominal surgery.

DETAILED DESCRIPTION:
Surgical factors that may affect the mobility of patients undergoing abdominal surgery should be examined, as well as individual characteristics and characteristics related to the postoperative period. If nurses know about the factors that may affect the patient's mobility after surgery, this may be helpful in effectively managing these factors in clinics and encouraging the patient to be more active.

This study was conducted to determine the mobility of patients who underwent abdominal surgery in the early postoperative period and the factors affecting mobility.

ELIGIBILITY:
Inclusion Criteria:

* • had no chronic pain or no visual or hearing impairment,

  * were 18 years of age or older,
  * were conscious after surgery,
  * had walked for the first time in the patient room after the surgery according to the clinical routine,
  * were voluntary to participate in the study.

Exclusion Criteria:

Fifty four patients who did not speak Turkish and 28 patients who failed to walk for the first time after surgery were excluded from the study.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The population of the study consisted of 236 patients who underwent cholecystectomy, appendectomy, hernia surgery and bariatric surgery in the general surgery clinic of the specified hospital on the dates of data collection. Among these patients, 152 patients who met the sampling criteria and volunteered to participate in the study were included in the sample.
Sampling Method: Non-Probability Sample
Enrollment: 152 (Actual)
Dates: Start 2019-09-01 (Actual); Primary Completion 2019-12-20 (Actual); Study Completion 2019-12-20 (Actual)

PRIMARY OUTCOMES:
Patient Mobility Scale | at day 1
  Through the patient mobility scale, the observer assesses the pain and difficulty experienced while exercising four activities in the postoperative period: "turning from one side of the bed to the other", "sitting on the edge of the bed", "standing up on the edge of the bed" and "walking in the patient room". The severity of perceived pain was rated on a five-point Likert-type scale anchored at "no pain(1)", " a little pain (2)", "moderate pain (3)", "a lot of pain (4)", "the worst pain (5)"; and the degree of difficulty was rated on a five-point Likert-type scale anchored at "very easy (1), easy (2), a bit difficult (3), difficult (4), and very difficult (5)" to determine how much pain and difficulty they felt. The pain and difficulty scores for each movement are summed up separately. The minimum and maximum scores for pain and difficulty are 4 and 20, respectively. A higher score means an increase in the degree of pain and difficulty of the movement.

SECONDARY OUTCOMES:
Observer Mobility Scale | at day 1
  This scale assesses the extent to which patients are dependent/independent during the movements, and the observer measures blood pressure, pulse rate and respiratory rate two minutes before and two minutes after the movement. Patients are assessed on a 1-5-point scale for their dependence while doing the movements. One point on the scale means that the patient can move independently, while five points means that the patient is unable to move despite verbal warnings and physical assistance. The total score of the scale is obtained by summing the scores for the four movements: "turning from one side of the bed to the other", "sitting on the edge of the bed", "standing up on the edge of the bed" and "walking in the patient room". The minimum and maximum scores of the scale are 4 and 20, respectively. The higher the score, the greater the dependency during the movement
Questionnaire for Factors Affecting Movement | at day 1
  The form included 17 questions on post-operative nausea-vomiting, sleep duration, presence of visitors, feeling weak, fear of falling, needing someone while moving, presence of someone to support while moving, fear of wounds to dehiscence while moving, suffering from stress due to surgery, use of the medical devices, pain, uncomfortable clothes and lack of information on how to move.

CONTACTS AND LOCATIONS:
Locations (1):
- Ebru Karaaslan, Şehitkamil, Gazi̇antep, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No